CLINICAL TRIAL: NCT01312337
Title: A Phase II Trial of Gefitinib Monotherapy in Pretreated Patients With Advanced Non-small Cell Lung Cancer Not Harboring Active EGFR Mutations
Brief Title: Iressa for EGFR Mutation Negative Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Myung-Ju Ahn / Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-07-252
Record Dates: First submitted 2011-02-21; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Nonsmall Cell Lung Cancer
Keywords: gefitinib; EGFR mutation negative; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iressa for EGFR wild group (Experimental): salvage Iressa therapy for patients with EGFR mutation negative NSCLC patients
  Interventions: Drug: salvage iressa

INTERVENTIONS:
Drug: salvage iressa — Iressa 250mg per day until progression

SUMMARY:
The investigators will examine efficacy and toxicity of gefitinib in Korean patients with EGFR wild tumors diagnosed with direct sequence test.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven NSCLC
* Ineligibile for curative treatment (namely, stage IIIb or IV)
* History of one to three prior systemic chemotherapy tumors without active EGFR mutations (exon 19 deletion, L858R mutation in exon 21)
* At least one lesion that was unidimensionally measurable by computed tomography (by RECIST 1.1)
* 18 years old or older
* Performance status ECOG 0-2
* Adequate organ function as evidenced by the following:

  * Absolute neutrophil count > 1.0 x 109/L
  * Platelets > 75 x 109/L
  * Total bilirubin ≤ 1.5 UNL
  * AST and/or ALT < 5 UNL
  * Creatinine clearance ≥ 45mL/min

Exclusion Criteria:

* Previous EGFR TKI therapy history
* Systemic anticancer therapy within the previous 3 weeks
* Other invasive malignancy within the past 2 years except non-melanoma skin cancer, in situ cervix cancer, or papillary thyroid cancer
* Other concurrent illness that would preclude study participation (severe heart disease)
* Other concurrent physical condition (e.g., infectious disease) that would preclude study participation
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
To determine disease control rate at 8 weeks will be 35% or higher in the the study group | 6 months after the enrollment of the last patients

SECONDARY OUTCOMES:
The number of patients who live longer than 6 months after enrollment | 6 months after the enrollment of the last patients

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea